CLINICAL TRIAL: NCT03263962
Title: Canrenone Effects on Cardiovascular Mortality in Patients With Congestive Heart Failure: the Coffee-it Study
Brief Title: Canrenone Effects on Cardiovascular Mortality in Patients With Congestive Heart Failure (the Coffee-it Study)
Acronym: THE COFFEE-IT
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, MD, PhD, FESC, University of Pavia
Other Study IDs: 20170016069
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Cardiac Heart Failure Patients
Keywords: CHF; Canrenone
MeSH Terms: interventions — Canrenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With canrenone: Patients with canrenone
  Interventions: Drug: Canrenone
- Without canrenone: Patients without canrenone

INTERVENTIONS:
Drug: Canrenone — Evaluation of canrenone therapy in patients with CHF
  Groups: With canrenone

SUMMARY:
To evaluate canrenone effects compared to other therapies on cardiovascular mortality in patients with congestive heart failure and preserved systolic function after 12 years of evaluation.

DETAILED DESCRIPTION:
The investigators will verify patients with cardiac heart failure (CHF) and preserved systolic function and each patient must have all clinical evaluation through basal measurements of blood pressure, heart rate, biochemical tests, and color Doppler echocardiographic parameters for at least 12 years.

The investigators will evaluate the effects of an aldosterone antagonist as canrenone compared to a group without canrenone and the investogators will verify how many patients reported cardiovascular mortality or will survive.

ELIGIBILITY:
Inclusion Criteria:

* patients with CHF
* preserved systolic function (FE ≥ 45%)

Exclusion Criteria:

* severe hypertension identified by blood pressure ≥180/110 mmHg
* patients with impaired systolic function (FE < 45%)
* history of active hepatitis or cirrhosis
* impaired renal function
* hyperpotassemia
* diabetes

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with CHF and preserved systolic function with or without an aldosterone antagonist as canrenone.
Sampling Method: Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Progression of CHF | 12 years
  Echocardiografic data
Haemodynamic data | 12 years
  Systolic blood pressure (SBP, Diastolic blood pressure (DBP), Heart rate (HR)
Metabolic data | 12 years
  fasting plasma glucose (FPG), total cholesterol (TC), HDL-cholesterol (HDL-C), triglycerides (Tg), LDL-cholesterol (LDL-C), lipoprotein (a) [Lp(a)],
Renal function | 12 years
  Sodium, Potassium, Creatinine, Uric acid
Endocrine data | 12 years
  Aldosterone, Plasma brain natriuretic peptide (BNP), Plasma renin activity (PRA)
Cardiovascular mortality | 12 years
  Register data
Survival | 12 years
  Register data

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No